CLINICAL TRIAL: NCT02598180
Title: Single Arm,Open Label Study, to Evaluate the Safety and Performance of VergenixTM Flowable Gel in Patients With Lower Limb Ulcers (CP-FG-001)
Brief Title: VergenixTM Flowable Gel in Patients With Lower Limb Ulcers
Acronym: CP-FG-001
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Collplant (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-FG-001
Record Dates: First submitted 2015-10-22; First posted 2015-11-05 (Estimated); Last update posted 2019-02-20 (Actual); Status verified 2019-02

CONDITIONS: Lower Limb Ulcers

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- VergenixTM Flowable Gel (Experimental): VergenixTM Flowable Gel
  Interventions: Device: VergenixTM Flowable Gel

INTERVENTIONS:
Device: VergenixTM Flowable Gel — The VergenixTM Flowable Gel is supplied as powder contained in a syringe that will be hydrated with saline.

SUMMARY:
Vergenix Flowable Gel is indicated for the management of acute and chronic wounds

DETAILED DESCRIPTION:
Vergenix™ Flowable Gel is an advanced wound care device primarily made of lyophilized Type I recombinant human Collagen (rhCollagen) . Vergenix Flowable Gel is supplied as a powder contained in a syringe that will be hydrated with saline, forming a gel. The Vergenix™ Flowable Gel provides a scaffold for cellular invasion and capillary growth. A secondary dressing to cover and secure the primary Vergenix™ Flowable Gel wound site followed by a final dressing application that will wrap the wound and surrounding area

ELIGIBILITY:
Inclusion Criteria:

Patient is 18 years of age or older.

2. Patient has one of the following difficult-to-treat chronic ulcers in the

lower limb:

2.1. Neuropathic lower limb ulcer

2.2. Venous lower limb ulcer

2.3. Post traumatic lower limb ulcer

2.4. Post operative lower limb ulcer

3. In case of Neuropathic foot grade according to University of Texas

Classification 1A

4. Wound area measurement ranging between 1-20cm2.

5. Ulcer defined as grade ≥E on the granulometer scale.

6. Willing to adhere to the proper off-loading device (off loading cast,

healing shoe) according to investigator recommendation.

7. Female patients must have a negative serum pregnancy test at

screening and be willing and able to use a medically acceptable

method of birth control or declare that they are abstaining from sexual

intercourse, from the screening visit through the study termination

visit or be surgically sterile (bilateral tubal ligation, bilateral

oophorectomy, or hysterectomy) or post-menopausal. Postmenopausal

women are defined as women with menstruation cessation for

12 consecutive months prior to signing of the informed consent form.

8. Ability and willingness to understand and comply with study

procedures and to give written informed consent prior to enrollment in

the study.

Exclusion Criteria:

1. Acute ulcer
2. Multiple Ulcers on the lower limb.
3. Clinical evidence of infection in the soft tissue, joint and/or bone

   (osteomyelitis) as presented in the physical examination.
4. The wound is penetrating into deep structures and involves bone,

   tendon or joint.
5. Wound has necrotic tissue.
6. Wound with sinus tracts.
7. HbA1c>12.
8. Patients with any other skin disorder unrelated to the ulcer that is

   presented in adjacent to the target wound.
9. Clinically significant arterial vascular disease with Ankle-Brachial Index (ABI) index <0.45

   if the peripheral pulse is not palpable, or flatted Pulse Volume Recording (PVR) in case of non

   palpable arteries.
10. Patient is receiving, or has received within one month prior to

    enrollment any treatment known to impair wound healing, including

    but not limited to:, immunosuppressive drugs, cytotoxic agents,

    radiation therapy and chemotherapy.
11. Has active malignant disease of any kind. A patient, who has had a

    malignant disease in the past, was treated and is currently disease-free

    for at least 5 years, may be considered for study entry.
12. Patients who present with significant metabolic co-morbidity that

    would preclude wound healing such as end stage renal failure, dialysis

    or severe liver dysfunction.
13. Clinically significant abnormalities in hematology and blood

    chemistry lab tests at screening that in the opinion of the investigator

    might interfere with the patient's safety or participation in the study.
14. Known positive HIV.
15. Known history of a significant medical disorder, which in the

    investigator's judgment contraindicates the patient's participation.
16. Known hypersensitivity and/or allergy to collagen.
17. Drug or alcohol abuse (by history).
18. Patients participating in any other clinical trials.
19. Patients with inability to communicate well with the investigators and

staff (i.e., language problem, poor mental development or impaired

cerebral function).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2014-11-25 (Actual); Primary Completion 2015-11-02 (Actual); Study Completion 2015-11-02 (Actual)

PRIMARY OUTCOMES:
Wound inspection | Change from baseline (day 0) to end of follow up (FU) period (week 4)
  Wound inspection is a combination of measures that includes assessing the wound grade (according to Texas classification for Neuropathic ulcers only), wound's area and depth, presence of granulation tissue and the percentage of wound area covered with granulation, quality of the granulation tissue (granulometer scale), presence and location of epithelialization, presence of necrotic tissue and percentage of wound area covered with necrotic tissue, amount and quality of wound's secretions, presence of infection.
Would Closure | Change from baseline (day 0) to end of follow up (FU) period (week 4)
Pain Assessment | Change from baseline (day 0) to end of follow up (FU) period (week 4)
  Pain will be assessed via VAS (Visual Analogue Scale) score
Blood Chemistry and Hematology | Change from baseline (day 0) to end of follow up (FU) period (week 4)
  The laboratory Blood Chemistry and Hematology tests will be aggregated to present the number of participants with abnormal laboratory values and/or Adverse Events that are related to treatment

SECONDARY OUTCOMES:
Adverse events | Change from baseline (day 0) to end of follow up (FU) period (week 4)
  Number of Participants With Adverse Events That Are Related to Treatment

CONTACTS AND LOCATIONS:
Overall Officials: Eran Tamir, MD, Principal Investigator — Maccabi Health Care
Locations (4):
- Israel (4):
  - Maccabi Health Care, Beersheba
  - Maccabi Health Care, Haifa
  - Maccabi Health Care, Tel Aviv
  - Assaf Harofeh, Zrifin